CLINICAL TRIAL: NCT00178360
Title: The Effects of Music Therapy on Depression, Chorea and Other Symptoms of Huntington's Disease
Brief Title: Effects of Music Therapy on Huntington's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, OJ Sahler, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10336
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease, Music Therapy, quality of life
MeSH Terms: conditions — Huntington Disease | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Therapy (Experimental): Subject will participate in one, individual, half-hour long music therapy session every other week and one hour-long group music therapy session each month, for a period of three months.
  Interventions: Behavioral: Music Therapy
- Standard Care (No Intervention): During the Standard Care time period, participants will continue to receive all of the medical care that they would normally receive for the treatment of Huntington's Disease, without the addition of music therapy services.

INTERVENTIONS:
Behavioral: Music Therapy — During individual Music Therapy sessions, subjects will participate in a variety of active music-making opportunities, including: playing musical instruments, singing, improvising, learning relaxation techniques, song writing, and/or lyric analysis. The activities for each session will be determined by both subject and therapist, and will be selected based on preference, emotional state, and desired goals for the day.
  Group music therapy sessions will focus on improving socialization, depression, and group dynamics. In this setting, the Music Therapist will choose from the following interventions:
  * Group singing
  * Group drumming
  * Music assisted relaxation
  * Group song writing
  * Lyric analysis
  * Improvisation
  * Music with art
  Arms: Music Therapy

SUMMARY:
The purpose of this study is primarily to assess the ability of a music therapy program to improve holistically the psychological, somatic, and social symptoms of patients with Huntington 's disease (HD). We hope to demonstrate the benefits of applying music therapy interventions to the management methods of HD, thus paving the way for the development of an effective music therapy program for individuals with HD.

DETAILED DESCRIPTION:
ABSTRACT

Background: Recent studies show that music therapy helps improve the symptomatic manifestations of Parkinson's Disease. Few studies have looked at music therapy as a treatment for the psychiatric, cognitive and motor symptoms of patients with Huntington's disease (HD).

Objective: To examine the feasibility and tolerability of a treatment program of music therapy for patients with Huntington's disease. Also, to determine if music therapy improves the mood and motor features of HD while improving quality of life.

Methods: Subjects with HD were recruited to participate in a six-week study that included one individual, half-hour music therapy session and one hour-long group session per week. The music therapy protocols were adapted from the Colorado State University's Neurological Music Therapy program and were targeted to HD symptoms including balance and posture, fine motor skills, memory and attention, vocalizations, and mood. In particular the protocols included Rhythmic Auditory Stimulation (RAS), Pattern Sensory Enhancement (PSE), and Therapeutic Instrumental Music Playing (TIMP). Primary outcome of tolerability was to be assessed by the subjects' adherence to the therapeutic protocol, attendance, and the results of an exit survey inquiring about their feelings toward the use of music therapy in HD. A secondary outcome of the study was the change in the Unified Huntington's Disease Rating Scale (UHDRS) score between baseline and study completion.

Results: Five subjects were recruited for study participation (one female and four males). Music therapy was found to be a tolerable and feasible treatment for patients with HD (100% adherence and 98% attendance). Exit surveys demonstrated strongly positive feelings towards the music therapy treatment program in four of the five subjects (one survey was completed with contradictory answers by the subject). While there was improvement in UHDRS scores for finger tapping, pronation/supination and the Luria, these changes did not achieve statistical significance with the small sample size in this study.

Conclusions: Music therapy was well tolerated among subjects with HD in this small study. Future studies are now being planned to look at the efficacy of this intervention in a larger population of HD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HD
* Over the age of 18
* Patients must be ambulatory, use of a walker or human support is acceptable
* Patients must be able to communicate their thoughts and feelings

Exclusion Criteria:

* Anyone without the preceding characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To examine the feasibility and tolerability of a treatment program of MT for subjects with HD. | End of Study

SECONDARY OUTCOMES:
To determine if MT improves the mood and motor features of HD while improving quality of life. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Frederick J Marshall, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Hyson C, Oliva R, LaDonna KA, Akwaa F, Richards J, Sahler OJ. "A Pilot Study of Music Therapy in Huntington' Disease". Journal of Neurology, Neurosurgery & Psychiatry 2005; 76:A29, Abstract P010.
- See also: American Music Therapy Association Home Page — http://www.musictherapy.org
- See also: Huntington's Disease Society of America Home Page — http://www.HDSA.org